CLINICAL TRIAL: NCT02927834
Title: The Role of Oral Steroids in the Management of Chronic Rhinosinusitis Without Nasal Polyps
Brief Title: Oral Steroids in Chronic Rhinosinusitis Without Nasal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Kristin Seiberling, MD, Principal Investigator, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5130196
Record Dates: First submitted 2016-08-04; First posted 2016-10-07 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Prednisone; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Antibiotic only (Active Comparator): 1. Augmentin (amoxicillin/clavulanate 875/125mg) orally (PO) twice a day for 3 weeks.
  Interventions: Drug: Augmentin
- Augmentin with 6 day steroid (Active Comparator): Augmentin with 6 day prednisone taper (40mg PO daily (QD) for 2 days, 20mg PO QD for 2 days, 10mg PO QD for 2 days, then stop)
  Interventions: Drug: 6 day Prednisone; Drug: Augmentin
- Augmentin with 21 day steroid (Active Comparator): Augmentin with 21 days prednisone taper (40mg PO QD for 5 days, 30mg PO QD for 5 days, 20mg PO QD for 5 days, 10mg PO QD for 5 days, then stop. )
  Interventions: Drug: Augmentin; Drug: 21 day Prednisone

INTERVENTIONS:
Drug: 6 day Prednisone — 6 day prednisone burst
  Arms: Augmentin with 6 day steroid
Drug: Augmentin — Antibiotic augmentin for 3 weeks
Drug: 21 day Prednisone — 21 day prednisone burst
  Arms: Augmentin with 21 day steroid

SUMMARY:
Chronic rhinosinusitis is a common disease that effects millions of people world wide. Despite its frequency it is unclear what treatment options are the best for these patients. Typically patients with chronic rhinosinusitis without nasal polyps (CRSsNP) are given a long term antibiotic (3 weeks), nasal steroid sprays, saline nasal irrigation and occasionally oral steroids. Oral steroids benefit patients with chronic rhinosinusitis with nasal polyps (CRSwNP) however their role in non polyp patients is less clear. It is the goal of this study to see if oral steroids benefit the treatment outcomes in those patients with chronic rhinosinusitis without nasal polyps. In addition this study will look to see if a short course (5 day burst) versus a longer course (21 day taper) of oral steroids make a difference in outcomes.

DETAILED DESCRIPTION:
The investigators will compare patients with CRSsNP who are treated with antibiotics/nasal steroid sprays, and compare them to chronic sinusitis patients who receive antibiotics/nasal steroid spray along with a course of oral steroids. The goal is to determine if oral steroids have a role in CRSsNP, and if so, the most effective dosage.

ELIGIBILITY:
Inclusion Criteria:

1. They have three-months of persistent symptoms meeting criteria for chronic rhinosinusitis as defined by the taskforce on rhinosinusitis.
2. They have a CT-scan in the clinic or have a viewable recent (< 3 weeks prior to clinic visit) CT-scan with a Lund Mackay score of 6 or greater. A Lund Mackay score of 6 or greater is felt to be indicative of at least moderate CRS.
3. They do not have nasal polyps on initial clinic nasal endoscopy
4. They are willing to participate in a clinical study
5. They are between the ages of 18 to 80.

Exclusion Criteria:

1. They have a condition in which the use of systemic corticosteroids is contraindicated such as diabetes will be excluded.
2. They are unable to or unwilling to take the prescribed antibiotics or steroids will excluded.
3. They have been treated with a > 3 week course of antibiotics and/or systemic steroids will also be excluded.
4. They have variants of chronic sinusitis known to be refractory to medical therapy such as Wegener's granulomatosis, primary ciliary dyskinesia or sarcoidosis.
5. They have sinusitis secondary to prior surgery, a dental procedure or anatomical variants.
6. They have nasal polyps on physical exam.
7. They are pregnant. Subjects who are possibly pregnant will be excluded based on history. Pregnancy testing is not standard of care for diagnostic imaging.
8. They have a Lund-Mackay score on CT scan of < 6
9. They are < 18 or > 80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antibiotic Only | Augmentin With 6 Day Steroid | Augmentin With 21 Day Steroid
Started | 8 | 8 | 8
Completed | 7 | 6 | 6
Not Completed | 1 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotic Only | Augmentin With 6 Day Steroid | Augmentin With 21 Day Steroid | Total
Number analyzed (Participants) | 7 | 6 | 6 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 5 | 14
  >=65 years | 2 | 2 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.28 (1) | 58.5 (1) | 41.2 (1) | 50.8 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 2 | 9
  Male | 5 | 1 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 5 | 5 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Sinonasal Outcome Test (SNOT 20)
Description: Sinonasal outcome test to access nasal/sinus symptoms. 20 questions, each question scored 0-5. 0 meaning no symptoms, 5 worse. 0- 100 total with lower number meaning better outcome
Time Frame: 4 weeks post treatment
Measure: Mean (95% Confidence Interval); unit: Score out of total 100
Arm/Group | Antibiotic Only | Augmentin With 6 Day Steroid | Augmentin With 21 Day Steroid
Number analyzed (Participants) | 7 | 6 | 6
Score out of total 100 | 50.33 [-2.21 to 56.29] | 53.14 [1.79 to 59.92] | 37 [2.85 to 39]

2. Primary Outcome: Nasal Endoscopy
Description: Physical exam findings of the nasal cavity. Scored 0-12. Lower score is better
Time Frame: 4 weeks post treatment
Measure: Mean (95% Confidence Interval); unit: score out of total 12
Arm/Group | Antibiotic Only | Augmentin With 6 Day Steroid | Augmentin With 21 Day Steroid
Number analyzed (Participants) | 7 | 6 | 6
score out of total 12 | 2.55 [-2.197 to 2.974] | 3.00 [1.793 to 3.492] | 2.16 [-2.37 to 3.37]

3. Primary Outcome: CT Scan Changes
Description: CT scan of the sinuses, Lund Mackay score to access severity of sinus disease on CT scan. Scored on scale 0-20 with lower score better.
Time Frame: 4 week post treatment
Measure: Mean (95% Confidence Interval); unit: score out of total 20
Arm/Group | Antibiotic Only | Augmentin With 6 Day Steroid | Augmentin With 21 Day Steroid
Number analyzed (Participants) | 7 | 6 | 6
score out of total 20 | 10.33 [8.15 to 11.3] | 11 [7.68 to 11.8] | 11.83 [5.13 to 13.15]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Patients were seen back in the office for adverse event collection
Arm/Group | Antibiotic Only | Augmentin With 6 Day Steroid | Augmentin With 21 Day Steroid
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT02927834/Prot_000.pdf